CLINICAL TRIAL: NCT00199758
Title: A Randomized Phase II Trial of Early Change of a Chemotherapeutic Doublet Versus Four Cycles of Chemotherapy in Advanced Non Small Cell Lung Cancer.
Brief Title: Study of an Early Change of a Chemotherapeutic Doublet Versus Four Cycles of Chemotherapy in Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I03022
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2007-11

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Non small cell lung carcinoma; Cisplatin; Gemcitabine; Paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: Gemcitabine
Drug: Taxol

SUMMARY:
The optimal strategy in advanced non small cell lung cancer with stable disease is not well known. There is no published study assessing an early change of chemotherapeutic drugs in these patients.Accordingly, we conduct this trial with the objective to improve the rate of objective responses by the switch to another doublet after 2 cycles of CDDP-gemcitabine association for patients with stable diseases (SD).

DETAILED DESCRIPTION:
Patients with stage IV NSCLC and measurable disease are included in a randomized phase II trial comparing for patients with stable disease after 2 cycles of a platin (P)-gemcitabine doublet (P d1: 75 mg/m2, gemcitabine 1 250 mg/m2 d1, d8 every three weeks) two subsequent cycles of this doublet (arm A) to a switch to another doublet (arm B) : paclitaxel 100 mg/m2 d1, d8, d15, gemcitabine 1 250 mg/m2 d1, d8, every four weeks.Platin, gemcitabine and paclitaxel are administered according nadir and pre-cycle haematologic evaluations (with dose decrease if needed). Response criteria are assessed with RECIST classification by the investigator panel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proved stage IV or pleural stage III NSCLC (neoplastic pleurisy confirmed).
* Metastatic relapses allowed in not irradiated area.
* Age between 18 and 70 years
* Chemonaïve patients
* At least one measurable target lesion according to recist criteria in non previously irradiated area.
* Performance status < 2
* Normal hepatic and renal function, absolute neutrophil count >1,5 giga/l, platelets >100 giga/l.
* Written informed consent.
* Life expectancy > 12 weeks.

Exclusion Criteria:

* SCLC, bronchial-alveolar and neuro-endocrine carcinoma.
* Previous chemotherapeutic treatment.
* Symptomatic brain metastases.
* Superior vena cava syndrome.
* Other concomitant diseases: heart failure, angina pectoris, arrhythmia , recent myocardial infarction.
* Peripheral neuropathy grade ≥2.
* Past or concomitance of another cancer except baso-cellular carcinoma of the skin or in situ cervical carcinoma.
* Hypersensitivity to paclitaxel or polysorbate 80.
* Pregnancy or breast feeding.
* Any concomitant radiotherapy, except palliative bone irradiation.
* Follow-up of the patient impossible.
* Prisoners.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227
Dates: Start 2003-09 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
1-Complete response
2-Partial response
3-Stable disease
4-Progression

SECONDARY OUTCOMES:
-Toxicity (NCI-CTC criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Vergnengre, MD, Principal Investigator — University Hospital, Limoges
Locations (21):
- France (21):
  - Service de Pneumologie, Beauvais
  - Service de Pneumologie, Bordeaux
  - Service de Pneumologie, Charleville Mezière
  - Service de Pneumologie, Créteil
  - Service de Pneumologie, Draguignan
  - Service de Pneumologie, Elbeuf
  - Service de Pneumologie, Gap
  - Service de Pathologie Respiratoire, Limoges
  - Service de Pneumologie, Hôpital de la Croix Rousse, Lyon
  - Service de Pneumologie, Mantes-la-Jolie
  - Département des Maladies Respiratoires, Marseille
  - Service de Pneumologie-Allergologie, Martigues
  - Service de Pneumologie, Meaux
  - Service de Pneumologie, Mulhouse
  - Service de Pneumologie - Hôpital St Antoine, Paris
  - Service de Pneumologie, Hôpital Pontchailloux, Rennes
  - Hôpital Charles Nicolle, Service de Pneumologie, Rouen
  - Service de Pneumologie, Hôpital Bois Guillaume, Rouen
  - Service de Pneumologie, Hôpital Nord, Saint-Etienne
  - Service de Pathologie Respiratoire, Toulon Naval
  - Service de Pneumologie, Villefranche

REFERENCES:
- [Background] Vergnenegre A, Tillon J, Corre R, Barlesi F, Berard H, Vernejoux JM, Le Caer H, Fournel P, Marin B, Chouaid C. A randomized phase II trial assessing in advanced non-small cell lung cancer patients with stable disease after two courses of cisplatin-gemcitabine an early modification of chemotherapy doublet with paclitaxel-gemcitabine versus continuation of cisplatin-gemcitabine chemotherapy (GFPC 03-01 Study). J Thorac Oncol. 2009 Mar;4(3):364-70. doi: 10.1097/JTO.0b013e318197f4ff. PMID 19155999